CLINICAL TRIAL: NCT05539417
Title: Snapshot Rectumcarcinoom 2016
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M. Kusters, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: 2020.366
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The treatment of rectal cancer is developing rapidly in the Netherlands, as well as internationally. This is accompanied by an increase in complexity of diagnosis and treatment, particularly when the tumor is located closer to the anorectal junction. Within these developments there is an important role for quality evaluation, where continuous feedback is able to improve care for rectal cancer in the Netherlands. By supplementing data from the Dutch ColoRectal Audit (DCRA) with additional data concerning diagnostics and treatment of rectal cancer patients operated in the year 2016, the Snapshot Rectumcarcinoom 2016 aimed to assess the improvement in surgical and oncological outcomes.

DETAILED DESCRIPTION:
Multiple changes in the treatment pathway for rectal cancer patients have contributed to the rapid developments over the last decade. First of all, in 2014 there has been revision of the guidelines, which adjusted MRI assessment and changed indications for neoadjuvant treatment. Moreover, the start of population screening has led to earlier detection of rectal cancer, which has increased attention for organ-sparing treatment. Furthermore, there has been a shift in surgical treatment towards more minimally invasive surgery and new techniques including robotic surgery and TaTME have been introduced. The centralization of care for rectal cancer patients has led to a decrease in number of hospitals that provide this care. These changes together ask for quality evaluation to provide feedback for further improvement of rectal cancer care in the Netherlands.

The Snapshot Rectumcarcinoom has been conducted retrospectively in 2021 concerning the patients operated in 2016 with a 4 year follow up. A similar snapshot study to evaluate outcomes of patients with rectal cancer who were operated in 2011 has been conducted retrospectively in 2015. This enables the Snapshot Rectumcarcinoom 2016 study to compare the oncological and surgical outcomes between 2011 and 2016.

Moreover, this study aimed to evaluate the practices and treatment of patients rectal cancer and enlarged lateral lymph nodes in 2016. Since the implementation of TME surgery there has been a shift toward more lateral recurrences, most likely caused by inadequate treatment of lateral lymph nodes. An international guideline for the appropriate treatment has been lacking, causing substantial variation practices. For example, lateral lymph nodes are often not mentioned by radiologists or during multidisciplinary meetings and there is no clear consensus concerning delineation of radiotherapy in lateral nodes. Moreover, in contrast to Asian countries, in the Netherlands surgical resection of the lateral lymphatic tissue is almost never done as clinicians have always relied on neoadjuvant treatment to sterilize the lateral compartment. Nevertheless, the Consortium study found that 16% of the population of rectal cancer patients had enlarged lateral lymph nodes, leading to a 19.5% 5-year lateral recurrence rate. When these nodes were removed by lateral lymph node dissection (LLND), this recurrence percentage was reduced to 5.7%. The Snapshot study aimed assess the current heterogeneity in diagnostics and treatment of lateral lymph nodes and increase awareness by training of the different specialties.

ELIGIBILITY:
Inclusion Criteria:

* Primary rectal cancer
* Operated in 2016 in a Dutch hospital
* Registred in the DCRA-register

Exclusion Criteria:

* Wait and see
* Resection for regrowth after wait and see

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent resection for primary rectal cancer in the Netherlands in 2016.
Sampling Method: Non-Probability Sample
Enrollment: 3107 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
How do different variables affect oncological and surgical outcomes? | 2016-2020
  This study will evaluate development between 2011 and 2016 by comparing this cohort to the Snapshot 2011 study.
The variation in treatment and awareness of lateral lymph nodes in patients with rectal cancer. | 2016-2020
  This study aims to assess the variation in treatment and the awareness of lateral lymph nodes in patients with rectal cancer. To increase awareness and improve current practices, MRI reassessment after training of radiologists will take place. Moreover, delineation training will be given to radiation oncologists. After these improvements in current practice, evaluation of this training will take place.

SECONDARY OUTCOMES:
Anastomotic leakage | 2016-2020
  Percentage of anastomotic leakage
Permanent stoma rate | 2016-2020
  Permanent stoma rate
Presence of presacral abscess | 2016-2020
  Presence of presacral abscess

IPD SHARING:
Plan to Share IPD: Yes
IPD data that underlie results in a publication can be made available upon reasonable request
Time Frame: Starting after initial publication of data
Access Criteria: Requests will be assessed by the study team

REFERENCES:
- [Result] Ogura A, Konishi T, Cunningham C, Garcia-Aguilar J, Iversen H, Toda S, Lee IK, Lee HX, Uehara K, Lee P, Putter H, van de Velde CJH, Beets GL, Rutten HJT, Kusters M; Lateral Node Study Consortium. Neoadjuvant (Chemo)radiotherapy With Total Mesorectal Excision Only Is Not Sufficient to Prevent Lateral Local Recurrence in Enlarged Nodes: Results of the Multicenter Lateral Node Study of Patients With Low cT3/4 Rectal Cancer. J Clin Oncol. 2019 Jan 1;37(1):33-43. doi: 10.1200/JCO.18.00032. Epub 2018 Nov 7. PMID 30403572
- [Result] Ogura A, Konishi T, Beets GL, Cunningham C, Garcia-Aguilar J, Iversen H, Toda S, Lee IK, Lee HX, Uehara K, Lee P, Putter H, van de Velde CJH, Rutten HJT, Tuynman JB, Kusters M; Lateral Node Study Consortium. Lateral Nodal Features on Restaging Magnetic Resonance Imaging Associated With Lateral Local Recurrence in Low Rectal Cancer After Neoadjuvant Chemoradiotherapy or Radiotherapy. JAMA Surg. 2019 Sep 1;154(9):e192172. doi: 10.1001/jamasurg.2019.2172. Epub 2019 Sep 18. PMID 31268504
- [Derived] van Geffen EGM, Verheij FS, Hazen SMJA, Sluckin TC, Consten ECJ, Dekker JT, Nederend J, Peeters KCMJ, de Wilt JHW, van Dieren S, Hompes R, Tuynman JB, Marijnen CAM, Tanis PJ, Kusters M; Dutch Snapshot Research Group. Oncological outcomes of planned and unplanned low Hartmann's procedure and restorative low anterior resection for rectal cancer: a population-based cross-sectional study. Tech Coloproctol. 2025 Nov 23;30(1):4. doi: 10.1007/s10151-025-03169-5. PMID 41276685
- [Derived] Moolenaar LR, van Geffen EGM, Hazen SJA, Sluckin TC, Beets GL, Leijtens JWA, Talsma AK, de Wilt JHW, Tanis PJ, Kusters M, Hompes R, Tuynman JB; Dutch Snapshot Research Group; Collaborators Snapshot Registry. Salvageable locoregional recurrence and stoma rate after local excision of pT1-2 rectal cancer - A nationwide cross-sectional cohort study. Eur J Surg Oncol. 2025 Jun;51(6):109623. doi: 10.1016/j.ejso.2025.109623. Epub 2025 Jan 23. PMID 40009914
- [Derived] Sluckin TC, Hazen SJA, Horsthuis K, Beets-Tan RGH, Antonisse IE, Berbee M, van Bockel LW, Boer AH, Ceha HM, Cnossen JS, Geijsen ED, den Hartogh MD, Hendriksen EM, Intven MPW, Leseman-Hoogenboom MM, Meijnen P, Muller K, Oppedijk V, Rozema T, Rutten H, Spruit PH, Stam TC, Velema LA, Verrijssen AE, Vos-Westerman J, Tanis PJ, Marijnen CAM, Kusters M; Dutch Snapshot Research Group. Coverage of Lateral Lymph Nodes in Rectal Cancer Patients with Routine Radiation Therapy Practice and Associated Locoregional Recurrence Rates. Int J Radiat Oncol Biol Phys. 2023 Oct 1;117(2):422-433. doi: 10.1016/j.ijrobp.2023.04.013. Epub 2023 Apr 28. PMID 37120027